CLINICAL TRIAL: NCT00281060
Title: Balloon Angioplasty Versus Stenting With Nitinol Stents in the Superficial Femoral Artery
Brief Title: Vienna Absolute Trial: Balloon Angioplasty Versus Stenting in the Superficial Femoral Artery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK164/2003
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2005-08

CONDITIONS: Atherosclerosis
Keywords: endovascular; balloon angioplasty; stents
MeSH Terms: conditions — Atherosclerosis

INTERVENTIONS:
Procedure: primary stenting

SUMMARY:
Minimal invasive treatment (called "endovascular") of the arteries of the lower limb remains problematic, because recurrent disease ("restenosis") frequently leads to recurrent symptoms. As yet, balloon angioplasty remains the recommended strategy to revascularize the superficial femoral artery (artery of the thigh). We investigated whether the use of a vascular endoprosthesis ("stent") improves patients´ outcome.

Study hypothesis: Primary stenting with self expanding nitinol stents may improve patency after endovascular treatment of superficial femoral artery obstructions compared to balloon angioplasty with optional stenting.

DETAILED DESCRIPTION:
STUDY DESIGN. From June 2003 to August 2004, we screened consecutive patients referred for endovascular treatment of the SFA due to intermittent claudication or chronic critical limb ischemia for enrollment in a randomized single-institution trial. Patients who were potential candidates for percutaneous intervention were discussed twice weekly in a consensus meeting of angiologists, vascular surgeons and interventional radiologists prior to being considered for trial enrollment. The protocol was approved by the institutional ethics committee, and patients provided written informed consent.

The clinical criterion for study entry was symptomatic peripheral artery disease (PAD) with either severe intermittent claudication (Rutherford class 3) or chronic critical limb ischemia with rest pain (Rutherford class 4) or ischemic ulcers (Rutherford class 5)1. Anatomic inclusion criteria, based upon findings on biplane DSA at the time of intervention, were a >50% stenosis or occlusion of the ipsilateral SFA with a target lesion length above 30mm, and at least one patent (<50% stenosis) tibio-peroneal run-off vessel. Exclusion criteria were acute critical limb ischemia, previous bypass surgery or stenting of the SFA, untreated inflow disease of the ipsilateral pelvic arteries (>50% stenosis or occlusion), and known intolerance of study medications or contrast agent.

STUDY END POINTS. The primary study end point was the binary rate of restenosis in the treated segment within 6 months postintervention by computed tomography angiography (CTA) or digital subtraction angiography (DSA). Restenosis was defined as a >50% lumen diameter reduction in the worst angiographic view at the most narrow site within the limits of the treated segment plus the adjacent ten millimeters proximal and distal to the treated segment.

Secondary end points were

1. anatomic outcome parameters: binary restenosis >50% by duplex ultrasonography (3, 6 and 12 months); angiographic degree of restenosis (% diameter reduction at 6 months); occurrence of stent fractures by biplane X-ray (6 and 12 months);
2. clinical outcome parameters: Rutherford stage of PAD and maximum walking capacity on the treadmill (24 hours, 3, 6 and 12 months); amputation and death (until 12 months);
3. hemodynamic outcome parameters: resting ankle brachial index (ABI) (24 hours, 3, 6 and 12 months).

Evaluation of all follow-up data and adjudication of primary and secondary end points were performed by two independent blinded observers. Discordances were resolved in consensus with a third blinded investigator.

INTERVENTIONS. Interventions were performed percutaneously from an antegrade or an over-the-bifurcation approach using 6 French sheaths. Biplane DSA was performed using two views at least 30° apart to evaluate lesion morphology, inflow disease and run-off. For precise documentation of the location of the lesion and the site of intervention a ruler was fixed at patients´ thigh with the distal end exactly overlapping the upper edge of the patella.

After successful wire passage through the target lesion, patients were randomly assigned to either primary stent implantation or PTA with optional secondary stenting, using computer generated random digits with randomization by blocks of four and sealed envelopes. Stratification criteria were claudication versus critical limb ischemia, and length of the target lesion (≤ versus > 60 mm).

In the stent group, primary stenting without predilation was performed except in patients with very tight stenoses or heavily calcified lesions that did not allow primary passage with the stent introducer device. Stents were implanted to extend 10 mm proximal and distal to the margins of the target lesion. When multiple stents were required, the margins of the stents were overlapped for 10 mm. Postdilation after stenting was performed strictly within the stented segment with up to 10% oversizing of the post-dilation balloon.

In the PTA group the minimal time for each balloon inflation was 2 minutes at 10 to 12 atmospheres. After dilation of the entire target segment, biplane control angiograms were obtained. In cases with a suboptimal primary result, defined as a residual stenosis >30% or presence of a flow limiting dissection in the worst angiographic view, a second prolonged balloon dilation (>2 minutes) of the target segment was performed. In patients with a persistent suboptimal result after the second balloon dilation, secondary stenting was performed.

For stent implantation in both groups, self-expandable nitinol stents (Dynalink / Absolute, Guidant, Santa Clara, CA) with a nominal diameter of 6 mm were used. Biplane angiograms were performed after the intervention in both treatment groups, using the same angles and magnifications as the baseline angiograms.

MEDICAL THERAPY. All patients received aspirin 100mg daily indefinitely and clopidogrel 75 mg daily for 3 months postintervention. Aspirin and clopidogrel were initiated at least 2 days prior to the intervention in most patients; otherwise a loading dose of 300 mg clopidogrel was given during the intervention.

SURVEILLANCE PROTOCOL. Examinations were performed at baseline and at 24 hours, 3 months, 6 months and 12 months after randomization, including staging of PAD by Rutherford1, measurement of resting ABI, treadmill exercise testing (3.2 km/h at 12° slope), and color duplex ultrasonography16. At 6 and 12 months X-rays in two planes were obtained for evaluation of stent fractures.

Angiographic evaluation of restenosis at 6 months was performed using either 16 slice CTA or conventional intra-arterial DSA. CTAs were performed on a "Somatom Sensation 16" 16-row, multi-slice CT scanner (Siemens Medical Systems, Erlangen, Germany). The accuracy and specificity of multi-slice CT with automated reconstruction has been reported to be comparable to intra-arterial DSA17-20. All patients with a suspected restenosis (>50%) by CTA underwent a conventional DSA with confirmation of the diagnosis. We performed DSA rather than CTA as the initial imaging procedure in patients with a planned ipsilateral or contralateral (re)intervention at the 6-month follow-up visit.

STATISTICAL METHODS AND SAMPLE SIZE CALCULATION. A sample size of 100 to 110 patients was estimated to be necessary assuming 6-month restenosis rates of 50% in the PTA group3 and 25% in the nitinol stent group11. A two-sided p-value of 0.05 was considered statistically significant and a power of 80% was required with a 10% maximum drop-out rate. Data analysis for primary and secondary study end points was performed according to the intention-to-treat principle. A secondary as-treated (per-protocol) analysis compared the results of stent implantation (primary or secondary) vs. PTA alone with respect to the primary study end point.

Descriptive data are given as means ± SD, or, for non-normal distributions or censored data sets, as medians with interquartile ranges (range from the 25th to the 75th percentile), and were analyzed by Mann Whitney U tests. Proportions were compared by Chi square statistics with Yates' correction or exact tests, as appropriate. Kappa statistics with 95% confidence intervals were used to assess agreement between angiography and duplex ultrasound. Multivariable logistic regression analysis was applied to assess the association between treatment and restenosis and to adjust for potentially confounding factors. We converted the odds ratios derived from the multivariate model to risk ratios (RR) with 95% confidence intervals (CI). Multiplicative interaction terms and log likelihood ratio tests were used to test for interactions. Calculations were performed using Stata release 8.0 (Stata Inc. College Station, TX, U.S.).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral artery disease Rutherford stages 3 to 5
* >50% stenosis of the ipsilateral superficial femoral artery
* Lesion length >30mm
* At least one patent crural run-off vessel,

Exclusion Criteria:

* Acute criticla limb ischemia
* Previous ipsilateral bypass surgery or ipsilateral SFA stenting
* Untreated inflow disease
* Known intolerance to clopidogrel, aspirin or radiocontrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2003-06; Study Completion 2005-08

PRIMARY OUTCOMES:
Angiographic restenosis at 6 months

SECONDARY OUTCOMES:
restenosis by duplex ultrasound at 3,6 and 12 months
walking distance on the treadmill at 3, 6 and 12 months
ankle brachial index at 3, 6 and 12 months
stent fractures at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schillinger, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Result] Schillinger M, Sabeti S, Loewe C, Dick P, Amighi J, Mlekusch W, Schlager O, Cejna M, Lammer J, Minar E. Balloon angioplasty versus implantation of nitinol stents in the superficial femoral artery. N Engl J Med. 2006 May 4;354(18):1879-88. doi: 10.1056/NEJMoa051303. PMID 16672699